CLINICAL TRIAL: NCT00202345
Title: Assessment of the Use of Intravenous Iron Sucrose to Maintain Haemoglobin Levels and Delay the Onset of Use of Erythropoietic Agents and/or Dialysis in Stage 3/4 Chronic Kidney Disease
Brief Title: Iron Sucrose in Stage 3/4 Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iron Sucrose 61864
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure; Anemia
Keywords: Creatinine Clearance; Hemoglobin; Iron sucrose; Oral iron therapy; Ferritin; Transferrin saturation; Iron
MeSH Terms: conditions — Renal Insufficiency; Anemia | interventions — Ferric Oxide, Saccharated

INTERVENTIONS:
Drug: Iron sucrose

SUMMARY:
One of the complications of late stage kidney disease is the development of a low red blood cell count (anaemia/low haemoglobin concentration). The Australian Commonwealth government limits funding of medications (called erythropoietic stimulating agents) to those patients who have already developed anaemia.

There is evidence supporting the beneficial effects of maintaining a higher haemoglobin in these patients. Higher haemoglobin can delay the onset of dialysis and reduce the development of heart enlargement. However, the administration of erythropoietic stimulating agents is not without risk, including a high financial burden, worsening of high blood pressure and a rare complication called pure red cell aplasia.

Previous studies have shown that patients with chronic kidney disease require additional iron to maintain the production of red blood cells. Thus it would be timely to determine if the administration of iron sucrose to these patients can maintain a near normal haemoglobin concentration, without the need to start an erythropoietic stimulating agent and possibly delaying dialysis.

Study Hypothesis: That administration of iron sucrose is superior to standard care in the prevention of anaemia in patients with stage 3 /4 kidney disease.

DETAILED DESCRIPTION:
Eligible patients will be approached. Those who agree to partake in the study will, after enrolment (including informed consent), be randomized to one of 2 groups.

Group A: To receive intravenous iron sucrose to maintain supra-physiological measures of iron status ) Group A will be targeted to have ferritin levels between 300 and 500µg/L and/or a transferrin saturation of between 25 and 50%. Between 100 and 200mg of intravenous iron sucrose will be administered by slow bolus injection one- to two-monthly to achieve these levels.

Oral iron will not be used routinely in this group.

Group B: Will have oral iron therapy if required to maintain ferritin levels between 100 and 150µg/L and/or transferrin saturations >20% but <25%. Patients in Group B who are unable to tolerate oral iron will be administered iron sucrose if necessary to maintain acceptable iron levels.

Patients in Group B will therefore differ from those in Group A (a) through the routine use of iron sucrose and (b) through the maintenance of different ferritin and transferrin saturation levels.

ELIGIBILITY:
Inclusion Criteria:

1. Initial Hb concentrations ≥ 110g/L (males and females)
2. Calculated GFR ≤ 35mL/min (≤ 50mL/min for diabetics)
3. Demonstration of a clinically significant rise in creatinine and/or a drop in Hb concentration in the previous 18 months. If such data are not available, the investigator will make a decision regarding eligibility based on the clinical circumstances.

Exclusion Criteria:

1. Age > 80
2. Pregnancy*
3. Unstable ischaemic heart disease*
4. Uncontrolled, severe, congestive cardiac failure
5. Haemochromatosis or iron overload* (ferritin >300µg/L and TSAT >25%)
6. Liver failure
7. Myelodysplastic syndromes or monoclonal gammopathies
8. Active malignancy or gastrointestinal bleeding*
9. Persistent sepsis* or significant chronic inflammation (CRP > 25)*
10. Iron deficiency* (Ferritin <30ug/L and Tsat <15%)or other haematinic disorder
11. Active and significant haemolysis*
12. Previous organ transplantation
13. Concurrent or significant past (>6 months) immuno-suppression
14. Adult polycystic kidney disease
15. Current use of an ESA
16. On dialysis *: patients can still be considered eligible after condition is reversed or treated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in Hb concentration at 12 months or termination (dialysis, commencement of an ESA). Minimum permitted enrolment is 6 months.

SECONDARY OUTCOMES:
The secondary endpoints will be the change in renal function (calculated creatinine clearance), the quality of life, the time taken to dialysis, the time from randomization to the requirement of an ESA and the number of hospitalization days.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P McMahon, MD, Principal Investigator — Melbourne Health
Locations (6):
- Australia (6):
  - Central Coast Health, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia